CLINICAL TRIAL: NCT05768945
Title: Data Analysis for Drug Repurposing for Effective Alzheimer's Medicines (DREAM)- Semaglutide v DPP4 Inhibitors
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Rutgers University (Other); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Rishi J. Desai, Assistant Professor of Medicine, Brigham and Women's Hospital
Other Study IDs: 2019P003607-14
Record Dates: First submitted 2023-03-03; First posted 2023-03-15 (Actual); Results first posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — semaglutide; Dipeptidyl-Peptidase IV Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Semaglutide: Exposure group
  Interventions: Drug: Semaglutide
- DPP4 inhibitors (sitagliptin, saxagliptin, linagliptin, and alogliptin): Reference group
  Interventions: Drug: DPP-4 inhibitor

INTERVENTIONS:
Drug: Semaglutide — Semaglutide claim is used as the exposure group.
  Groups: Semaglutide
Drug: DPP-4 inhibitor — DPP4 inhibitors (sitagliptin, saxagliptin, linagliptin, and alogliptin) claim is used as the reference group.
  Groups: DPP4 inhibitors (sitagliptin, saxagliptin, linagliptin, and alogliptin)

SUMMARY:
This study aims to evaluate the comparative risk of dementia/Alzheimer's disease onset between patients treated with medications that target specific metabolic pathways and patients treated with alternative medications for the same indication.

DETAILED DESCRIPTION:
This is a non-randomized, non-interventional study that is part of the DREAM Study of Brigham and Women's Hospital. DREAM is led by Dr. Madhav Thambisetty, MD, PhD, Chief of the Clinical and Translational Neuroscience Section, Laboratory of Behavioral Neuroscience, National Institute on Aging (NIA) intramural research program. This study aims to evaluate the comparative risk of dementia/Alzheimer's disease onset between patients treated with medications that target specific metabolic pathways and patients treated with alternative medications for the same indication using healthcare claims data.

ELIGIBILITY:
Please see https://drive.google.com/drive/folders/1VRjPaaelXFyBbA5gV6pwB_ijSIMyIJ4N?usp=share_link or Appendix A(https://drive.google.com/drive/folders/1OgKQlxsJi9UWRDd3Kbaux_8adngoSnZY?usp=sharing) for full code and algorithm definitions.

Medicare timeframe: 2008 to 2019 (end of data availability).

Inclusion Criteria:

* 1. Aged >/= 65 years on the index date
* 2. Enrollment in Medicare Part A, B, and D with no HMO coverage for 365 days prior to and including cohort entry date
* 3. Diagnosis code for type 2 diabetes measured 365 days prior to drug initiation

Exclusion Criteria:

* 1. Prior history of dementia measured anytime prior to cohort entry date
* 2. Prior history of nursing home admission in the 365 days prior to the cohort entry date
* 3. Prior use of any GLP receptor agonists (semaglutide, exenatide, liraglutide, albiglutide, dulaglutide, lixisenatide) or DPP4 inhibitors
* 4. Prior use of Semaglutide or DPP4 inhibitors concomitantly on index date

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: This study will employ a new user, active comparator, observational cohort study design comparing semaglutide v DPP4 inhibitors (sitagliptin, saxagliptin, linagliptin, and alogliptin). The patients will be required to have continuous enrollment during the baseline period of 365 days before initiation of study drugs (index date). Follow-up for the outcome (dementia) differs between analyses. Follow-up begins the day after drug initiation (analysis 1, 3, 4); 180 days after drug initiation (analysis 2).
Sampling Method: Non-Probability Sample
Enrollment: 742670 (Actual)
Dates: Start 2022-11-30 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Madhav Thambisetty, MD, PhD, Principal Investigator — National Institute on Aging (NIA)
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- DPP4 Inhibitors: Reference group
  DPP4 inhibitors (sitagliptin, saxagliptin, linagliptin, and alogliptin) claim is used as the reference group.
Period: Overall Study
Arm/Group | Semaglutide | DPP4 Inhibitors
Started | 9073 | 733597
Completed | 7129 | 7129
Not Completed | 1944 | 726468

BASELINE CHARACTERISTICS:
Population: Study cohort after 1:1 propensity score matching
Groups:
- Total: Total of all reporting groups
Arm/Group | Semaglutide | DPP4 Inhibitors (Sitagliptin, Saxagliptin, Linagliptin, and Alogliptin) | Total
Number analyzed (Participants) | 7129 | 7129 | 14258
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 7129 | 7129 | 14258
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.71 (4.52) | 70.70 (4.65) | 70.71 (4.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3406 | 3342 | 6748
  Male | 3723 | 3787 | 7510
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 5943 | 5968 | 11911
  Black | 547 | 531 | 1078
  Hispanic | 130 | 116 | 246
  Asian | 131 | 141 | 272
  North American Native | 44 | 44 | 88
  Other | 139 | 132 | 271
  Unknown | 195 | 197 | 392
Dementia risk factors [Count of Participants; unit: Participants]
  Anxiety | 1094 | 1073 | 2167
  Bipolar Disorder | 131 | 145 | 276
  Hypertension | 6650 | 6618 | 13268
  Coronary artery disease | 2527 | 2578 | 5105
  Obesity | 4005 | 4030 | 8035
  Schizophrenia | 15 | 20 | 35
  Depression | 1335 | 1362 | 2697

OUTCOME MEASURES:

1. Primary Outcome: Time to Dementia Onset
Description: Time to dementia onset, i.e., Alzheimer's disease, vascular dementia, senile, presenile, or unspecified dementia, or dementia in other diseases classified elsewhere. Please refer to uploaded protocol for full definition due to size limitations.
Time Frame: Median follow up times: 1) 98 days (exp), 134 days (ref) 2) 118 days (exp), 132 days (ref) 3) 90 days (exp), 308 days (ref) 4) 99 days (exp), 135 days (ref)
Population: Study cohort after 1:1 propensity score matching
Measure: Number (95% Confidence Interval); unit: Incidence rate per 1000 person year
Arm/Group | Semaglutide | DPP4 Inhibitors
Number analyzed (Participants) | 7129 | 7129
Incidence rate per 1000 person year
  Analysis 1 | 4.40 [2.27 to 7.68] | 6.06 [3.70 to 9.36]
  Analysis 2 | 4.69 [1.28 to 12.02] | 6.71 [2.70 to 13.83]
  Analysis 3 | 2.80 [0.34 to 10.13] | 10.24 [6.96 to 14.54]
  Analysis 4 | 0.37 [0.01 to 2.04] | 0.61 [0.07 to 2.19]

ADVERSE EVENTS:
Time Frame: 'As-treated' follow-up approach - Median follow-up days of 98 (for Semaglutide) and 134 (for DPP4 Inhibitors)
Description: Our study did not capture Serious Adverse Events.
Arm/Group | Semaglutide | DPP4 Inhibitors
All-Cause Mortality (participants affected / at risk) | 24/7129 | 44/7129
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/7129 | 0/7129

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-07): https://cdn.clinicaltrials.gov/large-docs/45/NCT05768945/Prot_SAP_000.pdf